CLINICAL TRIAL: NCT07025187
Title: the Effect of Integrated Neuomuscular Inhibition Technique on Adult Females With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Maram Karam Mohammed, Head of the department, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSIRB200-612
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): All patients will receive a traditional medical program by an experienced neurologist in the form of Muscle relaxants tizanidine ,4 mg to 32 mg, Three times a day.
  Interventions: Drug: Muscle relaxants tizanidine
- experimental group (Experimental): Patients in experimental group (B) will receive the same program as control group (A) plus the INIT for upper trapezius and suboccipital muscles. The INIT program will be administrated three times a week for one month.
  Interventions: Drug: Muscle relaxants tizanidine; Other: integrated neuromuscular inhibition technique

INTERVENTIONS:
Drug: Muscle relaxants tizanidine — All patients will receive a traditional medical program by an experienced neurologist in the form of Muscle relaxants tizanidine ,4 mg to 32 mg, Three times a day for one month .
Other: integrated neuromuscular inhibition technique — Patients in experimental group (B) will receive the same program as control group (A) plus the INIT for upper trapezius and suboccipital muscles. The INIT program will be administrated three times a week for one month .
  Other Names: INIT
  Arms: experimental group

SUMMARY:
The purpose of the current study is investigating the effect of integrated neuromuscular inhibition technique on adult females with cervicogenic headache.

Methods: Forty females with cervicogenic headache will be recruited. Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive a traditional medical treatment, but group (B) will receive additional integrated neuromuscular inhibition technique.

DETAILED DESCRIPTION:
Measurements will be taken for all participants before the start of treatment program then after the end of 4 weeks treatment program, then after another 4 weeks of follow up.all patients will be evaluated for headache pain intensity, cervicogenic headache frequency, cervicogenic headache duration, cervical range of motion in all directions, the isometric endurance capacity of sternocledomastoid and anterior scalene, kinesiophobia, neck disability, and headache impact test-6.

All patients will receive a traditional medical program by an experienced neurologist in the form of Muscle relaxants tizanidine ,4 mg to 32 mg, Three times a day.

Patients in experimental group (B) will receive the same program as control group (A) plus the INIT for upper trapezius and suboccipital muscles. The INIT program will be administrated three times a week for one month.

ELIGIBILITY:
Inclusion Criteria:

1 - A diagnosis of CGH will be made by an experienced neurologist as per the International Classification of Headache Disorders 3rd edition (ICHD-3) , but not including occipital nerve blockage 2-Additional inclusion criteria will include female patients aged> 18 years and<60 years.

3-headache intensity ≥ 3 on eleven-point numerical rating scale at enrolment. 4-at least three-month history of headache with a mean frequency of > 1/week. 5-hypomobility of the upper cervical spine (C0 to C3) on manual examination; and reproduction of the headache on palpation of the upper cervical spine (C0 to C3).

6-In addition, patients should exhibit active trigger points within the suboccipital, and upper trapezius muscles, ipsilaterally over the symptomatic side reproducing their headache symptoms .

Exclusion Criteria:

* Patients will be excluded if they have any of the following:

  1. cervical radiculopathy,
  2. history of neck, shoulder trauma or surgery,
  3. history of intervention for head or neck pain within the previous 3 months,
  4. A diagnosis of other types of headaches using the criteria of ICHD-3.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
headache pain intensity | Baseline, 4 weeks and 8 weeks .
  headache pain intensity measured by 11-Numerical rating scale. Primary outcome updated to headache intensity to better reflect the study objective.

SECONDARY OUTCOMES:
kinesiophobia | Baseline, 4 weeks and 8 weeks .
  kinesiophobia will be measured by Arabic Tampa scale
Isometric endurance capacity of sternocledomastoid and anterior scalene | Baseline, 4 weeks and 8 weeks .
  The isometric endurance capacity of the sternocleidomastoid and anterior scalene will be assessed using an isometric test.
the impact of headaches on patients' lives | Baseline, 4 weeks and 8 weeks .
  the impact of headaches on patients' lives measured by Arabic headache impact test-6.
neck disability | Baseline, 4 weeks and 8 weeks .
  the neck disability will be measured by Arabic neck disability index
headache frequency | Baseline, 4 weeks and 8 weeks
  Cervicogenic headache frequency, which is a self-administered outcome variable, will be identified by asking patients to enter their CGH pain experience in a medical logbook every evening to find the number of painful days in the last week, ranging from 0 to 7 days.
headache duration | Baseline, 4 weeks and 8 weeks .
  Headache duration will be measured as the total hours of headache in the last week.
cervical ROM in all directions | Baseline, 4 weeks and 8 weeks .
  Cervical right and left lateral flexion, extension, and flexion ROM will be measured using the iPhone clinometer application, whereas cervical right and left rotation ROM will be measured using the iPhone compass application.

CONTACTS AND LOCATIONS:
Locations (1):
- Khalid enb elwaleed polyclinic, Tanta, Algharbia, Egypt